CLINICAL TRIAL: NCT02567058
Title: Biomechanical and Ultrasonic Assessment of the Achilles Tendon in Vivo (MEDUSAA)
Acronym: MEDUSAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AORT 2011-FP / MEDUSAA
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Alterations of the Achilles Tendon
Keywords: Achilles tendon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3 groups of subjects (Experimental): 3 groups:
  * group I : healthy volunters
  * group II : patient with an immobilisation (between 1 and 2 months)
  * group III : patient with an antecedent of Achilles tendon breakage during the 10 past years
  Each group have the same interventions : ultrasound exam, IPAQ questionnaire
  Interventions: Device: Ultrasound exam; Behavioral: IPAQ questionnaire

INTERVENTIONS:
Device: Ultrasound exam — Ultrasound exam with :
  * 2 successions of 3 measures repeated for 2 visits (day 0 and day 21) for group I
  * 1 succession of 3 measures repeated for 4 visits (day 0, day 14, day 45, day 90)for group II
  * 1 succession of 3 measures for group III
  Other Names: Achillus; Ergometer
Behavioral: IPAQ questionnaire — IPAQ questionnaire

SUMMARY:
Among Musculoskeletal disorders (MSD) the rupture of the Achilles tendon is the most common. Up today, the mechanical and elastic properties of the Achilles tendon are still unknown, and that both in healthy subjects in pathology. The viscoelastic properties or dynamic mechanical properties are directly related to the tendon of the health status and its elongation capacity.

The laboratory UMR Inserm U930 - CNRS ERL 3106 in Tours has developed a non-invasive ultrasonic device, named Achillus, which, via an ultrasonic probe, allowing to access the viscoelastic properties of the tendon during the contraction of the sural triceps.

This is what we want to do in this first protocol: in vivo observation of the normal values and variations, looking for changes related to hyper solicitation and finally trying to highlight a tendon fragility parameter for patients who have experienced of a Achilles tendon rupture.

DETAILED DESCRIPTION:
Musculoskeletal disorders (MSD) are among the main causes of pain and disability in adults. Tendon disorders are an important part of MSD. Among them, the rupture of the Achilles tendon is the most common, with a prevalence of about 18 to 100000. The disorder mostly affects men between 30 and 50 years. Up today, the mechanical and elastic properties of the Achilles tendon are still unknown, and that both in healthy subjects in pathology. The viscoelastic properties or dynamic mechanical properties are directly related to the tendon of the health status and its elongation capacity. Additional tests that we have to explore the Achilles tendon are ultrasound and MRI. They bring mainly morphological information but can not demonstrate the mechanical properties of the tendon.

For this purpose, the laboratory UMR Inserm U930 - CNRS ERL 3106 in Tours has developed a non-invasive ultrasonic device, named Achillus, which, via an ultrasonic probe, allowing to access the viscoelastic properties of the tendon during the contraction of the sural triceps. It is therefore important in the exploratory work we propose to have a proven method of calibration of forces applied to the tendon, which is why an ergometer laboratory biomechanics and bioengineering at UT Compiègne is associated with our experiments.

No human study has yet been conducted to evaluate this method in medically relevant situations such as hyper solicitation and incorporated rupture.

This is what we want to do in this first protocol: in vivo observation of the normal values and variations, looking for changes related to hyper solicitation and finally trying to highlight a tendon fragility parameter for patients who have experienced of a Achilles tendon rupture.

ELIGIBILITY:
Inclusion Criteria:

Groupe I

* Male
* Between 18 and 60 years-old
* Informed consent form signed
* Affiliated to medical insurance

Groupe II

* Male
* Between 18 and 60 years-old
* Informed consent form signed
* Affiliated to medical insurance
* pathology of lower limb, from surgical treatment, and requiring an immobilization longer than one month and lower than two months, with discharge without support. Inclusion in the study will be done during within 48h from the onset of the immobilization

Groupe III

* Male
* Between 18 and 60 years-old
* Informed consent form signed
* Affiliated to medical insurance
* Antecedent of unilateral Achilles tendon breakage during the last 10 years (without breakage during the year previous the inclusion).

Exclusion Criteria:

Groupe I

* Know pathologies of collagen
* Antecedent of surgery on studied lower limb, located under the knee
* Pathology requiring a relief, a sport stoppage prescribed by a physician for a lower limb pathology during the last 12 months
* Muscular or neurologic pathology with impact on lower limbs
* Acute pathology able to compromise quality of the research (infectious, organic failure, pain …)
* Treatments able to affect the results of the research (myorelaxant, molecule changing the muscular tonus, quinolones …)
* Adult under guardianship
* Person under an exclusion period of other biomedical research

Groupe II

* Know pathologies of collagen
* Antecedent of surgery on studied lower limb, located under the knee
* Pathology requiring a relief, a sport stoppage prescribed by a physician for a lower limb pathology during the last 12 months
* Muscular or neurologic pathology with impact on healthy lower limb
* Acute pathology able to compromise quality of the research (infectious, organic failure, pain …)
* Treatments able to affect the results of the research (myorelaxant, molecule changing the muscular tonus, quinolones …)
* Adult under guardianship
* Person under an exclusion period of other biomedical research

Groupe III

* Know pathologies of collagen
* Antecedent of surgery on studied lower limb, located under the knee
* Pathology requiring a relief, a sport stoppage prescribed by a physician for a lower limb pathology during the last 12 months (including a controlateral Achilles tendon breakage)
* Muscular or neurologic pathology with impact on lower limbs
* Acute pathology able to compromise quality of the research (infectious, organic failure, pain …)
* Treatments able to affect the results of the research (myorelaxant, molecule changing the muscular tonus, quinolones …)
* Adult under guardianship
* Person under an exclusion period of other biomedical research

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2012-12; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measures of received signals of the ultrasound sensors and measures of applied strength on the pedal during | up to 3 months
  This is the measure of received signals of the ultrasound sensors and measures of applied strength on the pedal during plantar flexion efforts.
  Untreated data will be treated to extract this following parameters :
  * Control of rotational strengths couple applied by the participant
  * Simultaneous speed measure of lateral wave along the Achilles tendon The set oh these data will be got with an initial isometric effort at 20, 50, 80% of the de maximal voluntary muscle contraction previously measured

SECONDARY OUTCOMES:
score IPAQ questionnaire | up to 3 months
  Clinical parameter :score questionnaire of average physical activity of persons, determined by IPAQ questionnaire
Examination data | baseline
  Examination data : age, size, weight, laterality, smoking history
time of hyper stress | up to 3 months
  time of hyper stress

CONTACTS AND LOCATIONS:
Locations (1):
- Univesity Hospital of Tours, Tours, France